CLINICAL TRIAL: NCT01658085
Title: Harmonic FOCUS Versus Conventional Technique in Total Thyroidectomy for Benign Thyroid Disease. A Randomized, Prospective Study
Brief Title: Budget Impact of Harmonic FOCUS in Thyroidectomy
Acronym: TIME
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Pablo Moreno Llorente, Chief endocrine Surgery Unit, Hospital Universitari de Bellvitge
Other Study IDs: EO-0618
Record Dates: First submitted 2012-07-17; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Multinodular Goiter
Keywords: Thyroidectomy; Multinodular goiter; Harmonic Focus; budget impact; Harmonic scalpel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: HARMONIC FOCUS®: Total thyroidectomy (total bilateral extracapsular lobectomy) for Multinodular Goiter with HARMONIC FOCUS®
  Interventions: Device: HARMONIC FOCUS®
- Control group: ACE14S: Total thyroidectomy (total bilateral extracapsular lobectomy) for Multinodular Goiter with ACE14S
  Interventions: Device: ACE14S

INTERVENTIONS:
Device: ACE14S — Total thyroidectomy (total bilateral extracapsular lobectomy) for Multinodular Goiter with ACE14S
  Other Names: ACE® Curved Shears, Code: ACE14S (EES, Cincinnati, OH, USA)
  Groups: Control group: ACE14S
Device: HARMONIC FOCUS® — Total thyroidectomy (total bilateral extracapsular lobectomy) for Multinodular Goiter with HARMONIC FOCUS®
  Other Names: FOCUS Curved Shear, Code:FCS9 (EES, Cincinnati, OH, USA)
  Groups: Study group: HARMONIC FOCUS®

SUMMARY:
Study Design Multinodular Goiter (MNG) patients requiring surgery were referred to the Endocrine Surgery Unit.

Indirect laryngoscopy was routinely performed preoperatively to assess normal motility in vocal folds (VF). Ultrasounds (US) study was performed the month previous to surgery to evaluate thyroid volume. Eligible patients met the following criteria: to have MNG, age between 18 and 80 and consent to be included in the study. Exclusion criteria included previous neck surgery, vocal fold impairment, permanent or transitory NSAID or analgesic treatment, coagulation disorders and any cognitive impairment.

Eligible patients were proposed to enter a randomized study with 2 arms in which we compared the use of two harmonic scalpel devices: ACE14S and Harmonic Focus (Ethicon Endo-Surgery, Cincinnati, OH, USA).

The main endpoint was operative time. Secondary endpoints were total and relative (%) time of use of the device along thyroidectomy, recurrent laryngeal nerve (RLN) injury and hypocalcaemia (both persistent or temporary), number of ligatures, length of skin incision, postoperative pain according to a visual scale of pain, QOL after thyroidectomy (EuroQOL) and budget impact analysis.

All patients were operated on by 2 surgeons, one senior (responsible for the Endocrine Surgery Unit) and one junior under supervision.

Randomization Randomization was performed the same day of surgery at the OR by using a closed envelope. Patients were randomized to Group I (ACE14S) or Group II (HF) and allocated in a 1:1 proportion; they reminded blinded until the end of the study about the device used.

The haemostasis device was communicated to the surgeon previous to start surgery. Medical staff of the Endocrine Surgery Unit collected clinical data.

Surgical Technique Total thyroidectomy (TT), defined as total bilateral extracapsular lobectomy 9, was performed using HF or ACE14S for vessel division. Monopolar and bipolar forceps for cutting and coagulation were routinely used. Ties were used under surgeon's criteria according to size of the vessels and/or the need to obtain haemostasis in the vicinity of the RLN when bipolar forceps were not considered safe enough.

DETAILED DESCRIPTION:
OBJECTIVE:

To disclose the potential advantages and outcomes of the new Harmonic Focus (HF) device compared to Harmonic Scalpel ACE14S (ACE-14S) in benign thyroid surgery.

STUDY DESIGN:

Controlled randomized study.

METHODS:

Harmonic Focus was compared to former ACE14S device in patients undergoing total thyroidectomy for Multinodular Goiter. The primary endpoint was time of surgery. Secondary endpoints were time of use of the device, % of use along the procedure, number of ligatures, blood loss, hypocalcaemia, recurrent laryngeal nerve impairment, postoperative pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Multinodular goiter (MNG), age between 18 and 80 and consent to be included in the study

Exclusion Criteria:

* previous neck surgery
* vocal fold impairment
* permanent or transitory NSAID or analgesic treatment,
* coagulation disorders
* any cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients met the following criteria: to have MNG, age between 18 and 80 and consent to be included in the study.
  Eligible patients were proposed to enter a randomized study with 2 arms in which we compared the use of two harmonic scalpel devices: ACE14S and Harmonic Focus (Ethicon Endo-Surgery, Cincinnati, OH, USA).
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Operative time | Surgical time from skin incision to closure (about 70 minutes)
  Operative time was measured from skin incision to removal of thyroid gland. The percentage of time using the device along TT was calculated as follows: time of use of the device x 100/ operative time.

SECONDARY OUTCOMES:
Total and relative (%) time of use of the device along thyroidectomy | From skin incision to removal of thyroid gland (about 30 minutes)
  The percentage of time using the device along surgery was calculated as follows: time of use of the device x 100/ operative time.
Recurrent laryngeal nerve (RLN) injury | From surgery to 6 months
  Patients with laryngeal nerve injury were controlled monthly by indirect laryngoscopy till 6 months or healing.
hypocalcemia (both persistent or temporary) | Daily, from surgery to discharge (24h), or up to 6 months
  Temporary hypocalcemia was measured daily, from surgery to discharge.
  Persistent hypocalcemia was followed up as follows:
  * Non-complicated patients: one week and six months after the operation date.
  * Complicated patients: every month until cure or up to 6 months after surgery.
postoperative pain according to a visual scale of pain | From surgery to 7 days
  Pain evaluation was obtained at 24h and 7 days after surgery during postoperative control by using an analogue-visual scale reporting also the type of analgesic and the number of doses. If there was any complication (including reoperation) that increased hospital stay, pain evaluation was performed each 24h until discharge.
QOL after thyroidectomy (EuroQOL) | 1st and 7th postoperative day
  QOL was evaluated by completing EQ-5D questionnaire when patients were scheduled for the study (1st and 7th postoperative day)
Number of ligatures | Day of surgery
  Number of ligatures during the procedure was measured to determine if its reduction would imply less surgical time consumption
Length of skin incision | Day of surgery
  Measured at the end of the operation, once the skin was closured.
budget impact analysis | From surgery to discharge (24h)
  costs of total thyroidectomy (all of them according to the prices of our center) and deducting those time-dependent costs saved with the reduction of OR time. The following concepts were considered: personnel (with the same surgical team composition for both alternatives), anesthesia drugs, medical devices, overheads, repayment of the Harmonic generator, hospital stay and admission/discharge fees.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Moreno, MD, PhD, Principal Investigator — Hospital UIniversitari de Bellvitge
Locations (1):
- Hospital UIniversitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain